CLINICAL TRIAL: NCT00699127
Title: Dose Organizing the Information Given to Parents of NICU Infants Reduce Their Anxiety?
Brief Title: Organizing the Information Given to Parents of NICU Infants in Order to Reduce Their Anxiety
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: After a discussion, we decided to withdraw the study.
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Erez Nadir, MD, Hillel Yaffe medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HY-19-2008-CTIL
Record Dates: First submitted 2008-06-14; First posted 2008-06-17 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-07

CONDITIONS: Anxiety
Keywords: anxiety; parents; NICU; prematurity; Anxiety of parents to NICU infants
MeSH Terms: conditions — Anxiety Disorders; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The group that will have lecture of information regarding infants in NICU.
  Interventions: Behavioral: Lecture
- 2 (No Intervention): The group that will not have lecture of information regarding NICU hospitalization

INTERVENTIONS:
Behavioral: Lecture — Lecture of information regarding prematurity, NICU hospitalization, etc.
  Arms: 1

SUMMARY:
Being a parent to a premature infant in NICU is an anxious state. Parents ask a lot of questions, and look for information all the time. Organizing the information given to parents could reduce their anxiety. The parents will be divided into two groups: one group will get organized information, by a lecture at the first week of their infant's life, and the other group will not. Of course, questions will be answered all the time. The parents will answer a questionnaire on the first week of the infant's life, and on the last week, just before releasing the infant home.

DETAILED DESCRIPTION:
Being a parent to a premature infant in NICU is an anxious state. Parents ask a lot of questions, and look for information all the time. Organizing the information given to parents could reduce their anxiety. The parents will be divided into two groups: one group will get organized information, by a lecture at the first week of their infant's life, and the other group will not. Of course, questions will be answered all the time. The parents will answer a questionnaire on the first week of the infant's life, and on the last week, just before releasing the infant home.

ELIGIBILITY:
Inclusion Criteria:

* Parents to premature infants, after releasing the mother

Exclusion Criteria:

* Term infants
* Hospitalized mother

Max Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Difference between questionnaires at the first week and the last week to hospitalization. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Study Chair — Hillel Yaffe medical center, Hadera, Israel
Locations (1):
- Hillel Yaffe medical center, Hadera, Hadera, Israel